CLINICAL TRIAL: NCT02276144
Title: Investigation on the Frequency and Obstetric Significance of Metabolic Syndrome and Non-alcoholic Fatty Liver During Pregnancy
Brief Title: Metabolic Syndrome and Non-alcoholic Fatty Liver During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Fatty liver in pregnancy
Record Dates: First submitted 2014-10-10; First posted 2014-10-28 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2019-04

CONDITIONS: Fatty Liver; Gestational Diabetes
MeSH Terms: conditions — Fatty Liver; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum for lab tests
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Liver ultrasound — For evaluate whether fatty liver is exist or not

SUMMARY:
The aim of this study is to evaluate the prevalence of metabolic syndrome, liver function abnormality and non-alcoholic fatty liver disease in early pregnancy patients, and the risk of pregnancy complications.

DETAILED DESCRIPTION:
In cases in which metabolic syndrome and non-alcoholic fatty liver are risk factors of obstetric complications, such as gestational diabetes (GDM) or preeclampsia (PE), we are able to offer systematic clinical results from determining the independent risk factor and developing a predictable model. Recently, obstetric complications, especially GDM and PE, have increased due to the growth of elder pregnancy. In addition, as liver dysfunction has been known to be an independent risk factor of diabetes, cardiovascular disease, high blood pressure and renal dysfunction, its clinical importance has risen. Metabolic syndromes, such as obesity, hypertension, type II diabetes and abnormal lipid profile, have been known for its importance in development of non-alcoholic fatty liver disease. Considering abnormal liver function being an independent risk factor of diabetes, cardiovascular disease, high blood pressure and renal dysfunction in normal adult patients, we are able to predict that liver dysfunction might be a high risk factor of obstetric complications in pregnant women. In previous studies, the frequency of liver dysfunction in normal pregnant women was obtained.

The purpose of this current study was to investigate the prevalence of metabolic syndrome, abnormal liver function and non-alcoholic fatty liver in early pregnancy and the related risks of obstetric complications.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient clinic patients of Seoul National University Hospital, Seoul Metropolitan Government Boramae Medical Center, Incheon Seoul Woman Hospital
* Agree with this study
* Do not drink excess amount of alcohol for recent 2 years

Exclusion Criteria:

* Do not agree with this study
* Do not perform blood tests
* Have underlying hepatobiliary diseases
* Take medications which can cause liver abnormalities

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1st trimester pregnancy women with singleton
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2014-11; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Compare prevalence of obstetric complications between non-alcoholic fatty liver and normal pregnant women | From date of enrollment until the date of delivery, assessed up to 35wks
  Obstetrical complications include gestational diabetes, preeclampsia, etc Non-alcoholic fatty liver diagnosed by using liver ultrasound result of 1st trimester and blood test (AST, APT)

CONTACTS AND LOCATIONS:
Overall Officials: Joong Shin Park, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul Women's Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Goverment Seoul National University Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Zhang J, Suo Y, Wang L, Liu D, Jia Y, Fu Y, Fan W, Jiang Y. Association between atherogenic index of plasma and gestational diabetes mellitus: a prospective cohort study based on the Korean population. Cardiovasc Diabetol. 2024 Jul 5;23(1):237. doi: 10.1186/s12933-024-02341-9. PMID 38970008
- [Derived] Lee SM, Hwangbo S, Norwitz ER, Koo JN, Oh IH, Choi ES, Jung YM, Kim SM, Kim BJ, Kim SY, Kim GM, Kim W, Joo SK, Shin S, Park CW, Park T, Park JS. Nonalcoholic fatty liver disease and early prediction of gestational diabetes mellitus using machine learning methods. Clin Mol Hepatol. 2022 Jan;28(1):105-116. doi: 10.3350/cmh.2021.0174. Epub 2021 Oct 15. PMID 34649307